# Liposarcoma Clinical Trials: Investigating Engagement Patterns and Participation Trends Among Patients

An Informed Consent Form For Patients With Liposarcoma in Power Clinical Trial's Observational Study

Date: September 8, 2023

What Should You Know About This Informed Consent Form?

If you are tasked with completing this paper, it signals the potential of your participation in an observational clinical trial designed exclusively for those who suffer from liposarcoma. This paper is a thorough guide that reveals the study's main aims, elaborate execution strategy, and multiple ramifications, both good and potentially negative. Before making a decision, it is critical to investigate the specifics of your possible participation, and receiving advice from a reliable source can give vital views. If any of the material in this document appears confusing or if questions arise, please know that the researcher is accessible to give explanation.

# Exploring the Investigation's Aim

Liposarcoma is a type of cancer that develops in the soft tissues of the body, specifically in the fat cells. It is a rare form of cancer and accounts for a small percentage of all soft tissue sarcomas. Soft tissues include muscles, tendons, blood vessels, nerves, and fat, among others.

The treatment approach depends on the subtype and stage of the liposarcoma, as well as the individual's overall health. Early detection and treatment can improve outcomes, so anyone with concerning symptoms should seek medical attention promptly.

Liposarcoma is best managed by a team of healthcare professionals, including oncologists and surgeons, who specialize in treating sarcomas.

Clinical studies with a special emphasis on liposarcoma are critical in determining the safety and efficacy of new therapies for this illness. These trials are critical in establishing if new medicines outperform conventional treatments and offer strong evidence to support their widespread adoption.

This study is unusual in that it focuses on the experiences of people who have liposarcoma as they actively participate in a clinical trial incorporating medicinal therapies. The major focus is on closely examining trial completion rates and voluntary withdrawals among these individuals.

## Unveiling the Essence of Observational Studies

You will be immersed in an observational study by participating in this medical trial, a special feature of clinical research that is methodically constructed to gain insights from undisturbed observation of patients while keeping their care plans.

Researchers will just observe your trip, methodically measuring the consequences of your condition without making any changes. This particular trial design is critical in increasing our understanding of the intrinsic evolution of a certain medical illness and its consequences for persons who have it. By actively participating in this observational study, you become an important contributor to broadening the frontiers of medical knowledge and driving advances in the care delivered to those suffering from the same condition.

# Differentiating This Trial From Other Liposarcoma Clinical Trials

Understanding the distinctiveness of this research experiment is critical. It operates on an observational basis, suggesting that your participation will not include any particular therapies or interventions. Understanding the whole range of liposarcoma clinical trials, including interventional studies in which participants follow different treatment regimens, is critical.

Making an educated decision regarding your possible involvement in a clinical trial necessitates an active approach that includes research and comparison of various trials. Clinicaltrials.gov and other platforms provide a wealth of information about

<u>research relevant to liposarcoma</u>. Furthermore, Power's specialized web platform offers a complete list of ongoing <u>liposarcoma clinical trials</u> that are actively recruiting volunteers. You empower yourself to firmly design your participation decision by completing careful research and getting a complete awareness of various clinical trial types.

## Active Participation in Clinical Trial Surveys

We cordially invite you to actively contribute your experiences in the framework of this observational clinical investigation. This attempt necessitates the completion of questionnaires every two weeks, which will take roughly 20-30 minutes of your valuable time. Furthermore, we are fully prepared to conduct check-in calls at quarterly intervals, a practice that will continue during your participation in the trial.

To emphasize its significance, it is critical to clarify that your participation in the trial's survey phase is totally optional. You have the freedom to choose whether to answer certain questions or finish the full questionnaire. Furthermore, you have the freedom to discontinue your participation in the trial anytime you see fit. Recognizing that the decision to enroll in a clinical study is very personal, we are dedicated to providing the appropriate assistance. Your privacy and comfort are our unshakable values, and we are committed to respecting and supporting your decision-making process throughout the trial.

# Preserving the Privacy of Your Answers

Ensuring the complete privacy of your information is of utmost importance throughout the entirety of this clinical trial. To protect your anonymity, we kindly ask that you refrain from sharing any personal or identifiable information in your responses to the questionnaires. The committed research team is resolute in their dedication to enhancing the protection of your privacy. Nevertheless, it's important to acknowledge that certain legal situations may arise, necessitating the release of your data.

The total confidentiality of your information is critical for the duration of this research investigation. To safeguard your anonymity, we respectfully request that you abstain from including any personal or identifiable information in your questionnaire replies. The dedicated research team is steadfast in their commitment to improving the security of your privacy. Nonetheless, it is critical to recognize that some legal scenarios may occur that necessitate the sharing of personal data.

### Potential Health Risks

Despite the significant advances achieved by clinical trials, it is critical to recognize the possible health hazards that participants may face, particularly in studies evaluating novel medicines.

Nonetheless, our observational clinical research takes a unique strategy, purposefully minimizing these risks by foregoing the use of innovative therapies in individuals. Rather, our major focus is on rigorous monitoring and outcome evaluation in order to avoid any unnecessary health hazards.

### Possible Benefits

While immediate benefits may not be apparent for participants in this observational clinical research, their participation has the potential to influence others. The data collected from participants will be used to improve future techniques for enrolling liposarcoma individuals, potentially widening the scope of medical study. Individuals who embark on this therapeutic voyage have the ability to spark dramatic change within the area of medical research, potentially influencing the trajectory of future liposarcoma sufferers.

# Embarking on a Quest for Diversity in Clinical Trials

A plethora of internet resources await your active engagement if you are motivated by an insatiable curiosity to dig into the delicate realm of representation in clinical trials.

Whether your goal is to comprehend the complexities of the obstacles and possibilities associated with clinical trial diversity or to broaden your personal perspectives, the following resources might be invaluable:

Hussain-Gambles, Mahvash, Karl Atkin, and Brenda Leese. "Why ethnic minority groups are under-represented in clinical trials: a review of the literature." *Health & social care in the community* 12, no. 5 (2004): 382-388.

Huang, Xiaoli, Jimmy Lin, and Dina Demner-Fushman. "Evaluation of PICO as a knowledge representation for clinical questions." In *AMIA annual symposium* proceedings, vol. 2006, p. 359. American Medical Informatics Association, 2006.

# Confirmation of Informed Participation

I thus acknowledge that I have spent sufficient time understanding and internalizing the information included in the informed consent form, either by independent examination or with the assistance of a trusted individual who has expressed its essence to me. All of my concerns and anxieties have been thoroughly handled to my entire satisfaction.

I am fully aware that my participation in this study is the result of my personal decision, and I retain the only right to withdraw my consent without being required to offer justification or assume financial liabilities. It has been made clear to me that a copy of this informed consent form will be given for my own records.

After careful consideration and review of all of the material supplied to me, I hereby extend my approval to participate in this study, representing my informed and autonomous decision.

| Participant Name |
|-----------------------|
| Participant Signature |
| <br>Date |

Confirmation by Informed Consent Facilitator

I affirm that I have had a thorough conversation with the participant, meticulously unraveling the complexities encompassed in this written material. My goal was to ensure that the participant completely understood the research's main aims, methodology used, potential risks and benefits, and other critical components inherent to the liposarcoma clinical trial.

The participant was given ample opportunity, which encouraged the formation of questions and facilitated the explanation of concerns or misconceptions. It is critical to emphasize that the patient's participation in this study is the result of their voluntary decision, and they have the unfettered right to withdraw at any time, for any reason, without incurring any financial responsibilities.

Following the granting of consent by the participant, a meticulously kept duplicate of this written document was handed to them, functioning as a repository for their particular information.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |